CLINICAL TRIAL: NCT03058380
Title: Examining Stated-Preferences in Knee Arthroplasty: Unicompartmental Knee Arthroplasty (UKA) or Total Knee Arthroplasty (TKA)
Brief Title: Stated-Preferences in Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Duke Clinical Research Institute (Other); Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00079625
Record Dates: First submitted 2017-02-16; First posted 2017-02-20 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-05

CONDITIONS: Arthritis; Knee Osteoarthritis; Arthropathy of Knee
MeSH Terms: conditions — Arthritis; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stated-Preferences Evaluation Group: A stated-preferences evaluation instrument will be provided to participants with knee pain in the Stated-Preferences Evaluation Group. The instrument will measure patient preferences for total knee replacement versus unicompartmental knee replacement.
  Interventions: Other: Stated-Preferences Evaluation Instrument

INTERVENTIONS:
Other: Stated-Preferences Evaluation Instrument — A discrete choice experiment (Stated-Preferences Evaluation Instrument) will be electronically configured using best practice stated-preference methods to quantify preferences for total knee replacement versus unicompartmental knee replacement surgery.

SUMMARY:
The primary objectives of this study are to apply best-practice stated-preference methods to quantify patient preferences for benefit-risk tradeoffs associated with arthroplasty treatment options for end-stage osteoarthritis of the knee. Duke will develop and administer stated-preference surveys to adult patients (Ages 40-80) with knee pain to collect preference data, estimate the relative importance of treatment features and outcomes, and estimate maximum acceptable risks for given benefits and minimum acceptable benefits for given harms. This study proposal describes plans for the patient stated-preference survey.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80
* Knee Pain

Exclusion Criteria:

* Inability to read, understand and give effective English consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopaedic Clinics, Adult Reconstructive Surgery Clinics
Sampling Method: Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Patient Preference Measurements | 20 minutes
  Patient-stated preferences regarding treatment for knee pain based on questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Mather III, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No